CLINICAL TRIAL: NCT06067802
Title: A Phase II, Escalating Dose, Open Label Study to Evaluate the Safety of Triheptanoin for the Prevention of Hypoglycemia in Patients With Medium Chain Acyl-CoA Dehydrogenase Deficiency (MCADD)
Brief Title: Study of Triheptanoin for the Prevention of Hypoglycemia in Patients With Medium Chain Acyl-CoA Dehydrogenase Deficiency (MCADD)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been temporarily stopped until another study is completed. Data from the other study may inform changes to this study.
Sponsor: Jerry Vockley, MD, PhD (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Jerry Vockley, MD, PhD, Chief, Division of Genetic and Genomic Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23040121; UX007-IST237 (Other Grant/Funding Number: Ultragenyx Pharmaceutical Inc.)
Record Dates: First submitted 2023-08-10; First posted 2023-10-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Medium-chain Acyl-CoA Dehydrogenase Deficiency
Keywords: Medium-chain Acyl-CoA Dehydrogenase Deficiency
MeSH Terms: conditions — Medium chain acyl CoA dehydrogenase deficiency | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Triheptanoin (Experimental): Open label study
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Open-label design with doses of triheptanoin up to 1.0 gm/kg triheptanoin
  Other Names: Dojolvi

SUMMARY:
This is a medical research study to test a medication in adult patients with a disease called medium-chain acyl-CoA dehydrogenase deficiency (MCADD). The medication is triheptanoin, which is currently FDA approved for the treatment of Long-Chain Fatty Acid Oxidation Disorders. Previous research suggests that triheptanoin may also be effective in the treatment MCADD. This study will investigate the safety and efficacy (how well it works) of triheptanoin in patients with MCADD.

DETAILED DESCRIPTION:
Participation in the study will require three overnight admissions at the Clinical and Translational Research Center at the UPMC Children's Hospital of Pittsburgh (also called the PCTRC). The total length of the study is 10 weeks.

Subjects will have blood work and an intravenous access line (IV) placed for several blood draws during the visit. Subjects will begin fasting during the admission, which means they may consume only non-caloric fluids (water, unsweetened black coffee or tea, or sugar-free beverages). Bloodwork will be collected during the fast. Following the completion of the fast, the subject will eat a meal and will receive the study drug, triheptanoin. The total time of fasting will be up to 24 hours.

Dosing for this study will begin at 0.2 gm/kg/day up to a dose of 1.0 gm/kg/day. The dose will be increased gradually to avoid gastric upset. The dose should be divided into 3 or 4 daily doses and given with food or liquid. The dose can be decreased if a subject experiences any gastric upset that indicates that they cannot tolerate the higher dose.

Subjects will return two more times (at Weeks 5 and 9) to undergo the overnight admission and 24-hour fasting procedures outlined above. After the Week 9 admission they will no longer take the triheptanoin. Study staff will contact them by phone one week later (Week 10) to make sure they are not experiencing any adverse effects.

All study procedures will be done at no cost to the subjects.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of MCAD deficiency with molecular confirmation.
* Age criteria age ≥ 16 years
* Able to perform and comply with study activities including overnight admission to the research unit at UPMC Children's Hospital Pittsburgh, placement of an IV catheter, and all blood draws.
* Negative pregnancy test for all female subjects of child bearing age. Females of childbearning potential must agree to use a highly effective method of contraception, and males must agree not to father a child or donate sperm. True abstinence for the duration of the study will also be accepted.
* Signed informed consent for subjects ≥ 18 years, or assent by subjects age 16-17 years with parental consent for underaged subjects.

Exclusion Criteria:

* Use of any investigational drug within 30 days of screening.
* Active infection (viral or bacterial) or any other intercurrent condition as reported by the subject or noted on physical exam at screening.
* Evidence of liver disease as defined by elevations of AST or ALT> 1.5x ULN at screening
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at increased risk by participating in this study.
* Pregnant, planning to become pregnant, breastfeeding or lactating females.
* Diagnosis of pancreatic insufficiency or concomitant use of a pancreatic lipase inhibitor (e.g. Orlistat) which can interfere with absorption of triheptanoin
* Subjects with type 1 or type 2 diabetes, or who take medications as part of their routine care that can cause hypoglycemia

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE v5.0 | 10 weeks

SECONDARY OUTCOMES:
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C2 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C3 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C6 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C8 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C10 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C10:1 ratio levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C16 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in nmol/mL
Normalization of biochemical markers of disease (urine acylglycine) | 10 weeks
  Change in urine n-propionylglycine levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in mg/g creatinine
Normalization of biochemical markers of disease (urine acylglycine) | 10 weeks
  Change in urine suberylglycine levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in mg/g creatinine
Normalization of biochemical markers of disease (urine acylglycine) | 10 weeks
  Change in urine n-octanoylglycine levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in mg/g creatinine
Normalization of biochemical markers of disease (urine acylglycine) | 10 weeks
  Change in urine n-hexanoylglycine levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the number of participants who experience any change; measured in mg/g creatinine
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C2 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C3 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C6 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C8 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C10 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C10:1 ratio levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in nmol/mL
Normalization of biochemical markers of disease (plasma acylcarnitine) | 10 weeks
  Change in C16 levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in nmol/mL
Normalization of biochemical markers of disease (urine acylglycine) | 10 weeks
  Change in urine n-propionylglycine levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in mg/g creatinine
Normalization of biochemical markers of disease (urine acylglycine) | 10 weeks
  Change in urine suberylglycine levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in mg/g creatinine
Normalization of biochemical markers of disease (urine acylglycine) | 10 weeks
  Change in urine n-octanoylglycine levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in mg/g creatinine
Normalization of biochemical markers of disease (urine acylglycine) | 10 weeks
  Change in urine n-hexanoylglycine levels, comparing results from the fast before and after triheptanoin is initiated - this will be measured by the actual change from baseline to Week 10 for each participant; measured in mg/g creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Vockley, MD, PhD, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No